CLINICAL TRIAL: NCT05350553
Title: A Cross-Sectional Trial of Methylglyoxylated-Protein Levels in Adults With Chronic Pain
Brief Title: Methylglyoxal Evaluation in Humans
Acronym: MEH
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Doug Wright, Professor of Anatomy and Cell Biology, University of Kansas Medical Center
Other Study IDs: STUDY00148335
Record Dates: First submitted 2022-04-06; First posted 2022-04-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Neuropathy, Painful; Chronic Low-back Pain; Lumbar Disc Herniation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neuropathy, Painful; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Control: Patients 45-75 years of age without Type 2 Diabetes and without chronic low back pain.
- Type 2 Diabetic with Painful Neuropathy: Patients 45-75 years of age with Type 2 Diabetes and experiencing painful neuropathy (painful numbness or tingling in hands and/or feet)
- Chronic Low Back Pain as a Result of Lumber Disc Aberrancy: Patients 45-75 years of age with chronic low back pain as a direct result of non-operative lumber disc aberrancy (lumbar disc herniation, protrusion, or extrusion).

SUMMARY:
The investigators will test the hypothesis that patients with low back pain associated with lumbar disc aberrancy will have elevated MGO-protein levels circulating in the blood that are comparable to patients with painful diabetic neuropathy.

DETAILED DESCRIPTION:
This is a cross-sectional, non-interventional study conducted solely at KU Medical Center in which patients will be recruited and sorted based on the following status: 1) healthy, 2) painful diabetic neuropathy, 3) chronic low back pain as a result of non-operative lumbar aberrancy. Once recruited, subjects will undergo a venous blood draw to measure MGO-protein levels, HbA1c, blood glucose, NFL protein levels and GLO1 activity. Subjects will also complete questionnaires to better understand how MGO levels correlate with pain status.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the subject
* Able to read/speak English
* TYPE 2 DIABETES
* All healthy inclusion criteria AND
* Blood glucose levels > 126 mg/dl
* Diagnosed with neuropathy or experience painful numbness or tingling in their hands or feet
* LOW BACK PAIN
* All healthy inclusion criteria AND
* Chronic (persistent pain lasting longer than 3 months) low back pain as a direct result of non-operative lumbar disc aberrancy (disc herniation, protrusion, or extrusion)
* Aberrancy occurring within 12 months of pre-screening

Exclusion Criteria:

* Prisoner
* Current clinically significant cardiac or neurological disease
* Diagnosis of IBS, osteoarthritis, fibromyalgia, complex regional pain syndrome (CRPS), postherpetic neuralgia
* Lumbar surgery due to disc aberrancy
* Therapeutic spinal injections within the last 3 months (steroid, ablations, etc.)
* Chronic use of steroids or non
* steroidal anti-inflammatory drugs (NSAIDS) within 3 months of pre-screen
* Past or present use of spinal cord stimulators

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Based on their pain status, subjects will be distributed into three groups: healthy, type 2 diabetes with painful neuropathy, and chronic low back pain. Subjects will not be randomized as our studies are based on comparisons of subjects within the 3 groups. The study team will assess for the presence of neuropathy by verbal confirmation of the subject. Subjects placed within the chronic low back pain group must have a diagnosis of chronic pain symptoms (persistent pain lasting longer than 3 months), as a direct result of lumbar disc aberrancy in the last 12 months. The study team will require diagnostic imaging to confirm aberrancy status for enrollment in this group.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Methylglyoxal Evaluation | 12 months
  Number of participants with elevated blood methylglyoxal-derived hydroimidazolone (MG-H1, nM) with chronic pain.

SECONDARY OUTCOMES:
HbA1c | 12 months
  Quantify blood HbA1c.
Blood Glucose | 12 months
  Quantify non-fasting blood glucose (mg/dL).
Neurofilament Light | 12 months
  Quantify circulating neurofilament light (NFL, pg/mL) proteins.
Glyoxylase 1 Activity | 12 months
  Quantify glyoxylase 1 (GLO1, units) activity from blood cells.
Body Mass Index | 12 months
  Height (cm) and weight (kg) will be combined to report body mass index (kg/m^2).
Pain Status using the Brief Pain Index | 12 months
  Quantify patients' pain status using the Brief Pain Index (BPI).
Neuropathy Status using the Michigan Neuropathy Screening Index | 12 months
  Quantify patients' neuropathy status using the Michigan Neuropathy Screening Index (MNSI).

CONTACTS AND LOCATIONS:
Overall Officials: Doug Wright, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT05350553/ICF_000.pdf